CLINICAL TRIAL: NCT03345849
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Induction Study of the Efficacy and Safety of Upadacitinib (ABT-494) in Subjects With Moderately to Severely Active Crohn's Disease Who Have Inadequately Responded to or Are Intolerant to Conventional and/or Biologic Therapies
Brief Title: A Study of the Efficacy and Safety of Upadacitinib in Participants With Moderately to Severely Active Crohn's Disease Who Have Inadequately Responded to or Are Intolerant to Conventional and/or Biologic Therapies
Acronym: U-EXCEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-433; 2017-001240-35 (EudraCT Number)
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Results first posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-10

CONDITIONS: Crohn's Disease
Keywords: Upadacitinib; ABT-494; Efficacy; Safety; Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive placebo once daily for 12 weeks in Part 1. Clinical non-responders will receive 45 mg upadacitinib once daily for 12 weeks in Part 2.
  Interventions: Drug: Upadacitinib; Drug: Placebo for Upadacitinib
- Upadacitinib (Experimental): Participants will receive 45 mg upadacitinib once daily for 12 weeks in Part 1. Clinical non-responders will receive 30 mg upadacitinib once daily for 12 weeks in Part 2.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Oral; Tablet
  Other Names: ABT-494; RINVOQ
Drug: Placebo for Upadacitinib — Oral; Tablet
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of upadacitinib compared to placebo as induction therapy in adults with moderately and severely active Crohn's disease (CD).

DETAILED DESCRIPTION:
This study includes two parts:

* Part 1: a randomized double-blind placebo-controlled induction period and
* Part 2: an extended treatment period for non-responders from Part 1.

In Part 1, participants will be randomized in a 2:1 ratio to upadacitinib 45 mg once daily (QD) or matching placebo for 12 weeks. The randomization will be stratified by baseline corticosteroid use (yes or no), endoscopic disease severity (Simplified Endoscopic Score for Crohn's disease [SES-CD] < 15 and ≥ 15), and number of prior biologics with prior inadequate response or intolerance (0, 1, > 1).

Participants who do not achieve clinical response at Week 12 will be able to enroll in Part 2 to receive a double-blind extended treatment with upadacitinib until Week 24. Clinical response is defined as a ≥ 30% decrease in average daily very soft or liquid stool frequency (SF) and/or ≥ 30% decrease in average daily abdominal pain (AP) score (both not worse than Baseline).

Participants who achieve clinical response at Week 12 may be eligible to enter the 52-week, double-blind, maintenance portion of Study M14-430 (NCT03345823).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CD for at least 3 months prior to Baseline.
* Confirmed diagnosis of moderate to severe CD as assessed by stool frequency (SF), abdominal pain (AP) score.
* Evidence of mucosal inflammation based on the Simplified Endoscopic Score for Crohn's disease (SES-CD) on an endoscopy confirmed by a central reader.
* Demonstrated an inadequate response or intolerance to one or more conventional and/or biologic therapies (oral locally acting steroids, intravenous or oral corticosteroids, immunosuppressants or biologic therapies for CD), in the opinion of the investigator.

  * Note: Participants who have had inadequate response or intolerance to conventional therapy who have received prior biologic may be enrolled; however, participants must have discontinued the biologic for reasons other than inadequate response or intolerance (e.g., change of insurance, well controlled disease).
* If female, participant must meet the contraception recommendations.

Exclusion Criteria:

* Participant with a current diagnosis of ulcerative colitis or indeterminate colitis.
* Participant not on stable doses of CD related antibiotics, oral aminosalicylates, corticosteroids or methotrexate (MTX).
* Participant with the following ongoing known complications of CD: abscess (abdominal or peri-anal), symptomatic bowel strictures, fulminant colitis, toxic megacolon, > 2 entire missing segments of the following 5 segments: terminal ileum, right colon, transverse colon, sigmoid and left colon, and rectum, or any other manifestation that might require surgery while enrolled in the study.
* Participant with ostomy or ileoanal pouch.
* Participant diagnosed with conditions that could interfere with drug absorption including but not limited to short gut or short bowel syndrome.
* Screening laboratory and other analyses show abnormal results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (432):
- United States (119):
  - East View Medical Research, LLC /ID# 171176, Mobile, Alabama
  - CB Flock Research Corporation /ID# 166185, Mobile, Alabama
  - Delsol Research Management, Ll /Id# 170145, Chandler, Arizona
  - HonorHealth Research Institute - Shea /ID# 164821, Scottsdale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC /ID# 164803, Sun City, Arizona
  - Southern California Res. Ctr. /ID# 169655, Coronado, California
  - Citrus Valley Gastroenterology /ID# 166173, Covina, California
  - Hoag Memorial Hosp Presbyterian /ID# 222540, Irvine, California
  - United Medical Doctors /ID# 207449, Los Alamitos, California
  - Gastrointestinal Biosciences Clinical Trials, LLC /ID# 164762, Los Angeles, California
  - Facey Medical Foundation /ID# 203136, Mission Hills, California
  - United Medical Doctors - Murrieta /ID# 164945, Murrieta, California
  - Ucsd /Id# 164910, San Diego, California
  - Medical Assoc Research Grp /ID# 169706, San Diego, California
  - Univ of California San Francis /ID# 164944, San Francisco, California
  - Care Access Research /ID# 167767, San Pablo, California
  - Peak Gastroenterology Associates, PC /ID# 170143, Colorado Springs, Colorado
  - Delta Waves, Inc. /ID# 164776, Colorado Springs, Colorado
  - Western States Clinical Res /ID# 164760, Wheat Ridge, Colorado
  - Medical Research Center of CT /ID# 164926, Hamden, Connecticut
  - Clinical Research of West Florida, Inc /ID# 205827, Clearwater, Florida
  - Clinical Research of West Florida, Inc /ID# 208118, Clearwater, Florida
  - Advanced Research - Coral Springs /ID# 218021, Coral Springs, Florida
  - Encore Borland-Groover Clinical Research /Id# 203499, Jacksonville, Florida
  - Ctr for Advanced Gastroenterol /ID# 165353, Maitland, Florida
  - Crystal Pharmacology Research /ID# 166081, Miami, Florida
  - Coral Research Clinic /ID# 164890, Miami, Florida
  - Advanced Research Institute, Inc /ID# 164921, New Port Richey, Florida
  - Endoscopic Research, Inc. /ID# 206136, Orlando, Florida
  - Omega Research Maitland, LLC /ID# 203481, Orlando, Florida
  - Clinical Research Trials of Florida, Inc. /ID# 203485, Tampa, Florida
  - AdventHealth Tampa /ID# 171167, Tampa, Florida
  - Gastroenterology Associates of Central Georgia, LLC /ID# 165478, Macon, Georgia
  - Gastroenterology Consultants PC - Roswell /ID# 218220, Roswell, Georgia
  - Atlanta Gastroenterology Spec /ID# 164799, Suwanee, Georgia
  - Treasure Valley Medical Research /ID# 215032, Boise, Idaho
  - Rush University Medical Center /ID# 165497, Chicago, Illinois
  - University of Chicago Medicine /ID# 165503, Chicago, Illinois
  - DuPage Medical Group /ID# 205328, Downers Grove, Illinois
  - MediSphere Medical Research Center /ID# 166175, Evansville, Indiana
  - Indianapolis Gastroenterology /ID# 164938, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics /ID# 165436, Iowa City, Iowa
  - Tri-State Gastroenterology /ID# 165496, Crestview Hills, Kentucky
  - University of Louisville /ID# 165366, Louisville, Kentucky
  - University of Louisville /ID# 168572, Louisville, Kentucky
  - CroNOLA, LLC /ID# 164823, Houma, Louisiana
  - Nola Research Works, LLC /ID# 164759, New Orleans, Louisiana
  - Louisana Research Center, LLC /ID# 164894, Shreveport, Louisiana
  - Johns Hopkins University School of Medicine /ID# 211941, Baltimore, Maryland
  - MGG Group Co, Inc.Chevy Chase Clinical Research /ID# 164935, Chevy Chase, Maryland
  - Gastro Center of Maryland /ID# 171161, Columbia, Maryland
  - Lahey Hospital and Medical Center /ID# 214726, Burlington, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 164943, Ann Arbor, Michigan
  - Digestive Health Associates (DHA) - Farmington Hills /ID# 205793, Farmington Hills, Michigan
  - Center for Digestive Health /ID# 164822, Troy, Michigan
  - Clin Res Inst of Michigan, LLC /ID# 170133, Troy, Michigan
  - Mayo Clinic - Rochester /ID# 164783, Rochester, Minnesota
  - Southern Therapy and Advanced Research (STAR) LLC /ID# 165343, Jackson, Mississippi
  - Quality Clinical Research Inc. /ID# 170137, Omaha, Nebraska
  - Duplicate_CHI Nebraska d/b/a CHI Health /ID# 168578, Omaha, Nebraska
  - Las Vegas Medical Research /ID# 168588, Las Vegas, Nevada
  - AGA Clinical Research Associates, LLC /ID# 164769, Egg Harbor, New Jersey
  - Rutgers Robert Wood Johnson /ID# 166073, New Brunswick, New Jersey
  - NY Scientific /ID# 164931, Brooklyn, New York
  - United Health Services Hospitals, Inc /ID# 217485, Johnson City, New York
  - NYU Langone Long Island Clinical Research Associates /ID# 164927, Lake Success, New York
  - The Mount Sinai Hospital /ID# 170257, New York, New York
  - Columbia Univ Medical Center /ID# 164782, New York, New York
  - Gastoenterology Group of Rochester /ID# 166177, Rochester, New York
  - Richmond University Medical Center /ID# 201857, Staten Island, New York
  - Montefiore Medical Center - Moses Campus /ID# 166193, The Bronx, New York
  - Advantage Clinical Trials /ID# 168546, The Bronx, New York
  - Atrium Health Carolinas Medical Center /ID# 164932, Charlotte, North Carolina
  - PMG Research of Charlotte /ID# 171160, Charlotte, North Carolina
  - Wake Radiology UNC REX Healthcare - Raleigh Office /ID# 164904, Raleigh, North Carolina
  - Wake Forest Baptist Medical Center /ID# 164908, Winston-Salem, North Carolina
  - Plains Clinical Research Center, LLC /ID# 170140, Fargo, North Dakota
  - Gastro Health Research /ID# 164791, Cincinnati, Ohio
  - University of Cincinnati /ID# 164825, Cincinnati, Ohio
  - Cleveland Clinic Main Campus /ID# 209231, Cleveland, Ohio
  - The Ohio State University /ID# 170141, Columbus, Ohio
  - Optimed Research, Ltd. /ID# 205624, Columbus, Ohio
  - Hometown Urgent Care and Resea /ID# 201291, Dayton, Ohio
  - Dayton Gastroenterology, Inc. /ID# 167627, Englewood, Ohio
  - Great Lakes Medical Research, LLC /ID# 202010, Mentor, Ohio
  - Digestive Disease Specialists /ID# 201064, Oklahoma City, Oklahoma
  - Options Health Research, LLC /ID# 164820, Tulsa, Oklahoma
  - Healthcare Research Consultant /ID# 166195, Tulsa, Oklahoma
  - University of Pennsylvania /ID# 168430, Philadelphia, Pennsylvania
  - Pharmacorp Clinical Trials /ID# 164916, Charleston, South Carolina
  - Gastroenterology Associates, P.A. of Greenville /ID# 164771, Greenville, South Carolina
  - Rapid City Medical Center - GI Research /ID# 201735, Rapid City, South Dakota
  - Gastro One /ID# 164826, Germantown, Tennessee
  - East Tennessee Research Institute /ID# 203613, Johnson City, Tennessee
  - Quality Medical Research /ID# 205263, Nashville, Tennessee
  - Vanderbilt University Medical Center /ID# 164946, Nashville, Tennessee
  - TX Clinical Research Institute /ID# 164896, Arlington, Texas
  - Inquest Clinical Research /ID# 164785, Baytown, Texas
  - Texas Digestive Disease Consultants /ID# 209953, Cedar Park, Texas
  - Texas Digestive Disease Consultants /ID# 209801, Cedar Park, Texas
  - Baylor Scott & White Center for Inflammatory Bowel Diseases /ID# 170144, Dallas, Texas
  - CliniCore International, LLC /ID# 164902, Houston, Texas
  - Baylor College of Medicine - Baylor Medical Center /ID# 164947, Houston, Texas
  - Centex Studies, Inc. - Houston /ID# 201214, Houston, Texas
  - GI Specialists of Houston /ID# 202339, Houston, Texas
  - Caprock Gastro Research, LLC /ID# 215438, Lubbock, Texas
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 164786, San Antonio, Texas
  - Southern Star Research Institute, LLC /ID# 169755, San Antonio, Texas
  - Carl R. Meisner Medical Clinic /ID# 201061, Sugar Land, Texas
  - Tyler Research Institute, LLC /ID# 168687, Tyler, Texas
  - Gastro Health & Nutrition - Victoria /ID# 167812, Victoria, Texas
  - HP Clinical Research /ID# 164933, Bountiful, Utah
  - Advanced Research Institute /ID# 164784, Ogden, Utah
  - Duplicate_Care Access Research /ID# 164794, Salt Lake City, Utah
  - Velocity Clinical Research - Salt Lake City /ID# 166076, West Jordan, Utah
  - Washington Gastroenterology /ID# 164824, Bellevue, Washington
  - Virginia Mason Medical Center /ID# 164913, Seattle, Washington
  - The Vancouver Clinic, INC. PS /ID# 164918, Vancouver, Washington
  - Allegiance Research Specialists /ID# 165346, Wauwatosa, Wisconsin
- Argentina (6):
  - Cardio Alem /ID# 211285, San Isidro, Buenos Aires
  - Hospital Italiano de Buenos Aires /ID# 215541, Ciudad Autonoma Buenos Aires, Ciuadad Autonoma de Buenos Aires
  - Gedyt /ID# 210020, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Cemic /Id# 169182, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Hospital Provincial del Centenario /ID# 171252, Rosario, Santa Fe Province
  - Hospital Privado Univesitario /ID# 169230, Córdoba
- Australia (6):
  - Concord Repatriation General Hospital /ID# 171512, Concord, New South Wales
  - Coral Sea Clinical Research institute /ID# 212988, North Mackay, Queensland
  - Mater Misericordiae Limited /ID# 204909, South Brisbane, Queensland
  - Royal Adelaide Hospital /ID# 171514, Adelaide, South Australia
  - Box Hill Hospital /ID# 203736, Box Hill, Victoria
  - Fiona Stanley Hospital /ID# 171513, Murdoch, Western Australia
- Austria (2):
  - Medizinische Universitaet Wien /ID# 169465, Vienna, Vienna
  - Landeskrankenhaus Salzburg-Universitätsklinikum der PMU (LKH) /ID# 214470, Salzburg
- Belgium (3):
  - UCL Saint-Luc /ID# 200303, Woluwe-Saint-Lambert, Brussels Capital
  - CHU de Liege Sart Tilman /ID# 217534, Liège, Liege
  - AZ Sint-Lucas /ID# 200302, Ghent
- Bosnia and Herzegovina (4):
  - University Clinical Centre of the Republic of Srpska /ID# 208051, Banja Luka, Republika Srpska
  - University Clinical Center Tuzla /ID# 210325, Tuzla, Tuzlanski
  - Clinical Center University of Sarajevo /ID# 203887, Sarajevo
  - Polyclinic and Daily Hospital Dr. Al-Tawil /ID# 217842, Sarajevo
- Brazil (7):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva /ID# 166852, Goiânia, Goiás
  - Hospital Nossa Senhora das Graças /ID# 166863, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 166862, Porto Alegre, Rio Grande do Sul
  - Upeclin Fmb - Unesp /Id# 166867, Botucatu, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto - USP /ID# 166866, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC /ID# 208323, Santo André, São Paulo
  - Kaiser Clinica e Hospital Dia /ID# 166865, São José do Rio Preto, São Paulo
- Bulgaria (3):
  - UMHAT Kaspela EOOD /ID# 167613, Plovdiv
  - Duplicate_Second MHAT Sofia /ID# 167614, Sofia
  - MHAT Trakia /ID# 201679, Stara Zagora
- Canada (17):
  - University of Calgary /ID# 166974, Calgary, Alberta
  - Allen Whey Khye Lim Professional Corporation /ID# 168044, Edmonton, Alberta
  - University of Alberta - Zeidler Ledcor Centre /ID# 166971, Edmonton, Alberta
  - South Edmonton Gastroenterology Research Clinic /ID# 166978, Edmonton, Alberta
  - Fraser Clinical Trials Inc /ID# 166968, New Westminster, British Columbia
  - GIRI Gastrointestinal Research Institute /ID# 166975, Vancouver, British Columbia
  - QEII - Health Sciences Centre /ID# 169307, Halifax, Nova Scotia
  - Medicor Research Inc /ID# 166979, Greater Sudbury, Ontario
  - London Health Sciences Center /ID# 221038, London, Ontario
  - Scott Shulman Medicine Professional Corporation /ID# 169066, North Bay, Ontario
  - Taunton Surgical Centre /ID# 168043, Oshawa, Ontario
  - Ottawa Hospital Research Institute /ID# 212414, Ottawa, Ontario
  - Toronto Digestive Disease Asso /ID# 166972, Vaughan, Ontario
  - CISSS de Chaudière-Appalaches, Hôpital Hotel-Dieu de Lévis /ID# 166969, Lévis, Quebec
  - Centre Hospitalier de l'Universite de Montreal - CRCHUM /ID# 170120, Montreal, Quebec
  - Royal Victoria Hospital / McGill University Health Centre /ID# 170119, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS /ID# 170940, Sherbrooke, Quebec
- Chile (5):
  - M y F Estudios Clínicos /ID# 169984, Santiago, Region Metropolitana Santiago
  - Research Group /ID# 203179, Santiago, Santiago Metropolitan
  - Hospital Guillermo Grant Benavente de Concepción /ID# 212423, Concepción
  - CTR Estudios Clinicos /ID# 203941, Providencia
  - Hospital Clinico Universidad De Los Andes /ID# 207466, Santiago
- China (15):
  - Zhongshan Hospital Xiamen University /ID# 204984, Xiamen, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University /ID# 205228, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 204083, Guangzhou, Guangdong
  - The Sixth Affiliated Hosp Sun /ID# 204077, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 204081, Wuhan, Hubei
  - Nanjing Drum Tower Hospital /ID# 204900, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 204092, Nanchang, Jiangxi
  - The First Hospital of Jilin University /ID# 206868, Changchun, Jilin
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 204091, Shanghai, Shanghai Municipality
  - The second Affiliated hospital of Zhejiang University school of Medicine /ID# 204073, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital,Meical School Zhejiang University /ID# 204076, Hangzhou, Zhejiang
  - Beijing Friendship Hospital /ID# 204173, Beijing
  - The Second Xiangya Hospital of Central South University /ID# 204082, Changsha
  - Duplicate_Tianjin Med Univ General Hosp /ID# 206994, Tianjin
  - Tongji Hospital Tongji Medical College of HUST /ID# 204088, Wuhan
- Colombia (2):
  - Hospital Pablo Tobon Uribe /ID# 202404, Medellín, Antioquia
  - Hospital Universitario San Vic /ID# 200029, Medellín
- Croatia (6):
  - Clinical Hospital Dubrava /ID# 171185, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Sestre milosrdnice /ID# 205535, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 171203, Zagreb, City of Zagreb
  - Poliklinika Solmed /ID# 211519, Zagreb, City of Zagreb
  - UHC Split /ID# 171191, Split
  - Zadar General Hospital /ID# 205536, Zadar
- Czechia (4):
  - Nemocnice Ceske Budejovice a.s. /ID# 224389, České Budějovice
  - Hepato-Gastroenterologie HK, s.r.o. /ID# 171401, Hradec Králové
  - ARTROSCAN s.r.o. /ID# 200790, Ostrava
  - ResTrial s.r.o. /ID# 208653, Prague
- Denmark (4):
  - Herlev Hospital /ID# 202423, Herlev, Capital Region
  - Nordsjaellands Hospital /ID# 202424, Hilleroed, Capital Region
  - Kobenhavns Universitet - Hvidovre Hospital (HH) /ID# 202425, Hvidovre, Capital Region
  - Duplicate_Sjaellands Universitets Hospital /ID# 209445, Roskilde, Region Sjælland
- Egypt (6):
  - Clinical Research Center, Faculty of Medicine, Alexandria university. /ID# 171012, Alexandria
  - Clinical Research Center, Faculty of Medicine, Alexandria university. /ID# 171013, Alexandria
  - Clinical Research Center, Faculty of Medicine, Alexandria university. /ID# 209564, Alexandria
  - National Hepatology and Tropical Medicine Research Institute /ID# 170989, Cairo
  - Air Force Specialized Hospital /ID# 170996, Cairo
  - National Liver Institute /ID# 170988, Menoufiya
- West Tallinn Central Hospital /ID# 202785, Tallinn, Estonia
- France (3):
  - CHU Grenoble - Hopital Michallon /ID# 219034, La Tronche
  - Clinique Jules Verne /ID# 219073, Nantes
  - CH Valenciennes /ID# 219035, Valenciennes
- Germany (11):
  - Universitatsklinikum Mannheim /ID# 168759, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 203560, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 203552, Erlangen, Bavaria
  - Universitaetsklinikum Frankfurt /ID# 203566, Frankfurt am Main, Hesse
  - Zentrum für Gastroenterologie Saar MVZ GmbH /ID# 206741, Saarbrücken, Saarland
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 168757, Kiel, Schleswig-Holstein
  - Gastroenterologie am Mexikoplatz /ID# 203575, Berlin
  - Universitaetsmedizin Essen St. Josef Krankenhaus Werden /ID# 203570, Essen
  - Agaplesion Markus Krankenhaus /ID# 168758, Frankfurt am Main
  - Universitaetsklinikum Halle (Saale) /ID# 207455, Halle
  - Medizinisches Versorgungszentrum Portal 10 /ID# 200214, Münster
- Greece (5):
  - General Hospital of Athens Ippokratio /ID# 167045, Athens, Attica
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 202104, Athens, Attica
  - Tzaneio general hospital of Piraeus /ID# 206433, Piraeus, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 167044, Heraklion, Crete
  - General Hospital of Thessaloniki Hippokrateio /ID# 208825, Thessaloniki
- Tuen Mun Hospital /ID# 171218, Hong Kong, Hong Kong
- Hungary (11):
  - Mohacsi Korhaz /ID# 209441, Mohács, Baranya
  - CRU Hungary Egeszsegugyi és Szolgaltato Kft. /ID# 205547, Encs, Borsod-Abauj Zemplen county
  - Debreceni Egyetem Klinikai Kozpont /ID# 216419, Debrecen, Hajdú-Bihar
  - Bugat Pal Korhaz /ID# 201893, Gyöngyös, Heves County
  - Szent Borbala Korhaz /ID# 209897, Tatabánya, Komárom-Esztergom
  - Obudai Egeszsegugyi Centrum Kft. /ID# 201892, Budapest, Pest County
  - Semmelweis Egyetem /ID# 210167, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont /ID# 201724, Budapest
  - Debreceni Egyetem Kenezy Gyula Egyetemi Korhaz /ID# 201723, Debrecen
  - Pest Megyei Flor Ferenc Korhaz /ID# 206154, Kistarcsa
  - Mentahaz Maganorvosi Kozpont /ID# 201895, Székesfehérvár
- Mercy University Hospital /ID# 206511, Cork, Ireland
- Israel (6):
  - Soroka University Medical Center /ID# 169913, Beersheba, Southern District
  - Tel Aviv Sourasky Medical Center /ID# 204877, Tel Aviv, Tel Aviv
  - Assaf Harofeh Medical Center /ID# 204872, Be’er Ya‘aqov
  - Hadassah Medical Center-Hebrew University /ID# 169928, Jerusalem
  - Rabin Medical Center /ID# 202636, Petah Tikva
  - Kaplan Medical Center /ID# 170276, Rehovot
- Italy (14):
  - Policlinico Universitario Campus Bio-Medico /ID# 168183, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini /ID# 168184, Rome, Lazio
  - Istituto Clinico Humanitas /ID# 168185, Rozzano, Milano
  - Fondazione PTV Policlinico Tor Vergata /ID# 168188, Rome, Roma
  - Presidio Columbus-Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Un /ID# 168182, Rome, Roma
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 168186, Negrar, Verona
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna /ID# 168187, Bologna
  - A.O. Per L'Emergenza Cannizzaro /ID# 168190, Catania
  - Policlinico San Martino/Univer /ID# 168191, Genova
  - ASST Fatebenefratelli Sacco - Ospedale Fatebenefratelli e Oftalmico /ID# 168181, Milan
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 170849, Milan
  - Azienda Ospedaliero-Universitaria di Modena /ID# 201897, Modena
  - A.O. Ospedali Riuniti Villa Sofia - Cervello /ID# 168189, Palermo
  - Azienda Ospedaliero Universitaria Pisana-Stabilimento di Cisanello /ID# 202421, Pisa
- Japan (50):
  - Aichi Medical University Hospital /ID# 165971, Nagakute-shi, Aichi-ken
  - Nagoya University Hospital /ID# 165969, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 165970, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital /ID# 200175, Toyohashi, Aichi-ken
  - National Hospital Organization Hirosaki General Medical Center /ID# 165961, Hirosaki-shi, Aomori
  - Toho University Sakura Medical Center /ID# 165963, Sakura-shi, Chiba
  - Fukuoka University Chikushi Hospital /ID# 214404, Chikushino-shi, Fukuoka
  - Kurume University Hospital /ID# 166012, Kurume-shi, Fukuoka
  - National Hospital Organization Takasaki General Medical Center /ID# 167127, Takasaki-shi, Gunma
  - NHO Fukuyama Medical Center /ID# 167131, Fukuyama-shi, Hiroshima
  - Hiroshima University Hospital /ID# 166014, Hiroshima, Hiroshima
  - Asahikawa Medical University Hospital /ID# 167120, Asahikawa-shi, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 165960, Sapporo, Hokkaido
  - Sapporo Medical University Hospital /ID# 167124, Sapporo, Hokkaido
  - Sapporo IBD Clinic /ID# 223561, Sapporo, Hokkaido
  - Aoyama Clinic /ID# 166009, Kobe, Hyōgo
  - Hyogo College of Medicine College Hospital /Id# 165973, Nishinomiya-shi, Hyōgo
  - Kanazawa University Hospital /ID# 169218, Kanazawa, Ishikawa-ken
  - Iwate Medical University Uchimaru Medical Center /ID# 202464, Morioka, Iwate
  - Imamura General Hospital /ID# 227137, Kagoshima, Kagoshima-ken
  - Idzuro Imamura Hospital /ID# 206654, Kagoshima, Kagoshima-ken
  - Sameshima Hospital /ID# 206675, Kagoshima, Kagoshima-ken
  - Yokohama City University Medical Center /ID# 167128, Yokohama, Kanagawa
  - Japanese Red Cross Kyoto Daiichi Hosital /ID# 165972, Kyoto, Kyoto
  - Kyoto University Hospital /ID# 169889, Kyoto, Kyoto
  - Yokkaichi Hazu Medical Center /ID# 167196, Yokkaichi-shi, Mie-ken
  - Tohoku University Hospital /ID# 167122, Sendai, Miyagi
  - Nara Medical University Hospital /ID# 169219, Kashihara-shi, Nara
  - Kenseikai Dongo Hospital /ID# 208104, Yamatotakada-shi, Nara
  - Niigata University Medical & Dental Hospital /ID# 170045, Niigata, Niigata
  - Ishida Clinic of IBD and Gastroenterology /ID# 167121, Ōita, Oita Prefecture
  - Chikuba Hospital for Proctological and Gastrointestinal Diseases /ID# 166010, Kurashiki-shi, Okayama-ken
  - Okayama University Hospital /ID# 167356, Okayama, Okayama-ken
  - Kinshukai Infusion Clinic /ID# 218872, Osaka, Osaka
  - Osaka Metropolitan University Hospital /ID# 166015, Osaka, Osaka
  - Osaka University Hospital /ID# 169663, Suita-shi, Osaka
  - Osaka Medical and Pharmaceutical University Hospital /ID# 206326, Takatsuki-shi, Osaka
  - Tokitokai Tokito clinic /ID# 165962, Saitama-shi, Saitama
  - Shiga University of Medical Science Hospital /ID# 167129, Ōtsu, Shiga
  - Hamamatsu University Hospital /ID# 224352, Hamamatsu, Shizuoka
  - NHO Shizuoka Medical Center /ID# 167125, Sunto-gun, Shizuoka
  - Tokyo Medical And Dental University Hospital /ID# 165965, Bunkyo-ku, Tokyo
  - Tokai University Hachioji Hospital /ID# 165967, Hachioji-shi, Tokyo
  - The Jikei University Hospital /ID# 167130, Minato-ku, Tokyo
  - Kyorin University Hospital /ID# 165966, Mitaka-shi, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 205980, Shinjuku-ku, Tokyo
  - Toyama Prefectural Central Hospital /ID# 217834, Toyama, Toyama
  - Japanese Red Cross Wakayama Medical Center /ID# 200643, Wakayama, Wakayama
  - Wakayama Medical University Hospital /ID# 169482, Wakayama, Wakayama
  - Yamagata University Hospital /ID# 200157, Yamagata, Yamagata
- Latvia (3):
  - VCA Polyclinic Aura /ID# 169498, Riga
  - Pauls Stradins Clinical University Hospital /ID# 169519, Riga
  - Digestive Disease Center Gastro /ID# 169508, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 206936, Kaunas
  - Vilnius University Hospital Santaros Klinikos /ID# 203286, Vilnius
- Malaysia (3):
  - Hospital Sultanah Bahiyah /ID# 202626, Alor Star, Kedah
  - Universiti Sains Malaysia /ID# 200102, Kelantan, Kelantan
  - Universiti Kebangsaan Malaysia (UKM) Medical Centre /ID# 170773, Kuala Lumpur, Selangor
- Mexico (3):
  - Instituto de Investigaciones Aplicadas a la Neurociencias A.C. /ID# 207579, Durango, Durango
  - Morales Vargas Centro de Investigacion S.C. /ID# 203494, León, Guanajuato
  - Clinica de Investigacion en Reumatologia y Obesidad S.C. /ID# 207238, Guadalajara, Jalisco
- Netherlands (5):
  - Radboud Universitair Medisch Centrum /ID# 166928, Nijmegen, Gelderland
  - Zuyderland Medisch Centrum /ID# 169700, Heerlen, Limburg
  - Onze Lieve Vrouwe Gasthuis /ID# 166929, Amsterdam
  - Academisch Medisch Centrum /ID# 166927, Amsterdam
  - Medisch Spectrum Twente /ID# 170298, Enschede
- Poland (5):
  - Malopolskie Centrum Kliniczne /ID# 202167, Krakow, Lesser Poland Voivodeship
  - Vistamed /ID# 208572, Wroclaw, Lower Silesian Voivodeship
  - Centrum Zdrowia MDM /ID# 200491, Warsaw, Masovian Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkus /ID# 224301, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Reuma Park /ID# 200490, Warsaw, Masovian Voivodeship
- Portugal (5):
  - Hospital da Senhora da Oliveira Guimaraes, EPE /ID# 170245, Guimarães, Braga District
  - Hospital Egas Moniz /ID# 170253, Lisbon, Porto District
  - Unidade Local de Saúde do Alto Minho, EPE - Hospital Conde de Bertiandos /ID# 200607, Ponte de Lima, Viana do Castelo District
  - Hospital Garcia de Orta, EPE /ID# 170241, Almada
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 170248, Porto
- Puerto Rico (2):
  - Mindful Medical Research /ID# 203358, San Juan
  - School of Medicine University of Puerto Rico-Medical Science Campus /ID# 166771, San Juan
- Romania (3):
  - Institutul Clinic Fundeni /ID# 167817, Sector 2, București
  - Clinica GASTRO MED SRL /ID# 206369, Cluj-Napoca, Cluj
  - Cabinet Particular Policlinic Algomed /ID# 167818, Timișoara
- Russia (12):
  - Immanuel Kant Baltic Federal University /ID# 203811, Kaliningrad, Kaliningrad Oblast
  - LLC Medical Center /ID# 209236, Novosibirsk, Novosibirsk Oblast
  - Perm Clinical Center of the Federal Medical and Biological Agency /ID# 202990, Perm, Permskiy Kray
  - LLC Novaya Klinika /ID# 206616, Pyatigorsk, Stavropol Kray
  - Professor Pasechnikov Gastroenterology and Pankreatology clinic /ID# 202997, Stavropol, Stavropol Kray
  - Kazan State Medical University /ID# 169638, Kazan', Tatarstan, Respublika
  - Olla-Med Clinic /ID# 208720, Moscow
  - P.A. Bayandin Murmansk Regiona /ID# 169639, Murmansk
  - Republican hospital named after V.A. Baranov /ID# 206488, Petrozavodsk
  - Euromedservice /ID# 206610, Pushkin
  - X7 Clinical Research Center /ID# 216350, Saint Petersburg
  - City Clinical Hospital No. 31 /ID# 208868, Saint Petersburg
- Serbia (6):
  - Clinical Hosp Center Zvezdara /ID# 168214, Belgrade, Beograd
  - Military Medical Academy /ID# 168783, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 168215, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 168750, Belgrade, Beograd
  - University Clinical Center Kragujevac /ID# 205859, Kragujevac, Sumadijski Okrug
  - Clinical Center Vojvodina /ID# 168213, Novi Sad, Vojvodina
- Singapore (3):
  - KL Ling Gastroenterology and Liver Clinic /ID# 217962, Singapore
  - Gleneagles Medical Centre /ID# 206531, Singapore
  - Tan Tock Seng Hospital /ID# 203160, Singapore
- Slovakia (2):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 169958, Banská Bystrica
  - KM Management, spol. s.r.o. /ID# 170201, Nitra
- Univ Medical Ctr Ljubljana /ID# 217795, Ljubljana, Slovenia
- South Africa (6):
  - Farmovs (Pty) Ltd /Id# 207535, Bloemfontein, Free State
  - Lenasia Clinical Trial Centre /ID# 205145, Johannesburg, Gauteng
  - Wits Clinical Research Site /ID# 170852, Johannesburg, Gauteng
  - Allergy & Immunology (AIU) /ID# 171431, Cape Town, Western Cape
  - Dr JP Wright /ID# 170887, Cape Town, Western Cape
  - Private Practice Dr MN Rajabally /ID# 169853, Cape Town, Western Cape
- South Korea (10):
  - Hayang University GuriHospital /ID# 167587, Guri-si, Gyeonggido
  - CHA University Bundang Medical Center /ID# 167592, Seongnam-si, Gyeonggido
  - Kangbuk Samsung Hospital /ID# 167586, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 167590, Seoul, Seoul Teugbyeolsi
  - Inje University Haeundae Hospital /ID# 202630, Busan
  - Dong-A University Hospital /ID# 167591, Busan
  - Pusan National University Hospital /ID# 167589, Busan
  - Kyungpook National University Hospital /ID# 207019, Daegu
  - Samsung Medical Center /ID# 167588, Seoul
  - Chung-Ang University Hostipal /ID# 207018, Seoul
- Spain (11):
  - Hospital Universitari Son Espases /ID# 201998, Palma de Mallorca, Balearic Islands
  - Hospital Universitario de Navarra /ID# 202355, Pamplona, Navarre
  - Hospital Universitario A Coruna - CHUAC /ID# 203910, A Coruña
  - Hospital Clinic de Barcelona /ID# 201990, Barcelona
  - Hospital Universitario de Girona Doctor Josep Trueta /ID# 202645, Girona
  - Hospital Juan Ramon Jimenez /ID# 201995, Huelva
  - Hospital Universitario La Paz /ID# 201994, Madrid
  - Hospital Universitario de Salamanca /ID# 206358, Salamanca
  - Hospital Universitario Virgen Macarena /ID# 201993, Seville
  - Hospital Clinico Universitario de Valencia /ID# 209657, Valencia
  - Hospital Universitario y Politecnico La Fe /ID# 201992, Valencia
- Sweden (5):
  - Hallands Hospital Halmstad /ID# 170828, Halmstad, Halland County
  - Karolinska University Hospital Solna /ID# 224488, Solna, Stockholm County
  - Alingsas lasarett /ID# 170826, Alingsås, Västra Götaland County
  - Sodra Alvsborgs sjukhus /ID# 203077, Borås, Västra Götaland County
  - Sahlgrenska University Hospital /ID# 169171, Gothenburg, Västra Götaland County
- Switzerland (2):
  - Universitätsspital Zürich /ID# 170998, Zurich, Canton of Zurich
  - Inselspital, Universitätsspital Bern /ID# 170997, Bern
- Taiwan (3):
  - China Medical University Hospital /ID# 169791, Taichung
  - Taichung Veterans General Hospital /ID# 169790, Taichung
  - National Taiwan University Hospital /ID# 169792, Taipei
- Turkey (Türkiye) (10):
  - Acibadem Kozyatagi Hospital /ID# 209406, Kadıköy, Istanbul
  - Erciyes University Medical Fac /ID# 171331, Melikgazi, Kayseri
  - Ankara Univ Medical Faculty /ID# 206409, Ankara
  - Inonu Universitesi Turgut Ozal /ID# 201268, Battalgazi/malatya
  - Mustafa Kemal University Medic /ID# 171336, Hatay
  - Istanbul University Istanbul Medical Faculty /ID# 171364, Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi /ID# 171332, Istanbul
  - Mersin University Medical /ID# 171338, Mersin
  - Sisli Etfal Train & Res Hosp /ID# 171334, Şişli
  - Gazi Universitesi Tip Fakultes /ID# 217444, Yenimahalle
- Ukraine (6):
  - Medical Centre of "Ukrainian German Antiulcer Gastroenterology Centre BYK-KYIV" /ID# 203738, Kyiv, Kyivska Oblast
  - Kharkiv City Clinical Hospital No.2 n.a. Prof. O.O. Shalimov /ID# 167907, Kharkiv
  - Kyiv Municipal Clinical Hospital #18 /ID# 207889, Kyiv
  - MNI KRC Kyiv Regional Clinical Hospital /ID# 202454, Kyiv
  - Lviv Railway Clinical Hospital of branch Healthcare Centers of Public Joint Stoc /ID# 167908, Lviv
  - CNE Vinnytsya Regional Clinical Hospital named after N.I.Pirogov /ID# 222110, Vinnytsia
- United Kingdom (12):
  - South Eastern Health and Social Care Trust /ID# 205323, Belfast, Antrim
  - Warrington and Halton Hospitals NHS Foundation Trust /ID# 171383, Warrington, Cheshire West And Chester
  - Warrington and Halton Hospitals NHS Foundation Trust /ID# 209086, Warrington, Cheshire West And Chester
  - Royal United Hospitals Bath /ID# 169074, Bath
  - University Hospitals Birmingham NHS Foundation Trust /ID# 169070, Birmingham
  - The Dudley Group NHS Foundation Trust /ID# 169069, Dudley
  - King's College Hospital NHS Foundation Trust /ID# 169072, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 169075, Newcastle upon Tyne
  - Stockport NHS foundation trust /ID# 208719, Stockport
  - Taunton and Somerset NHS Foundation Trust /ID# 209665, Taunton
  - St George's University Hospitals NHS Foundation Trust /ID# 205552, Tooting
  - The Royal Wolverhampton NHS Trust /ID# 171382, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Vermeire S, Colombel JF, Danese S, Panaccione R, Peyrin-Biroulet L, Beck K, Chaparro M, Gisbert JP, Dubcenco E, Klaff J, Naling G, Ford S, Remple V, Joshi N, Suravaram S, Duncan B, Wang Y, Wick-Urban B, Loftus EV. Benefit-risk profile of upadacitinib: exploratory post hoc analysis of phase 2b/3 studies in patients with moderately to severely active ulcerative colitis or Crohn's disease. J Crohns Colitis. 2026 Jan 9;20(1):jjaf198. doi: 10.1093/ecco-jcc/jjaf198. PMID 41264726
- [Derived] Dubinsky MC, D'Haens G, Dewit O, Juillerat P, Panaccione R, Fujii T, Dubcenco E, Lacerda AP, Anyanwu SI, Ford S, Cunneen C, Fish I, Joshi N, Garrison A, Loftus EV. Efficacy and Safety with Upadacitinib by Baseline Corticosteroid Use in Patients with Moderately to Severely Active Crohn's Disease. Inflamm Bowel Dis. 2025 Nov 4:izaf250. doi: 10.1093/ibd/izaf250. Online ahead of print. PMID 41189093
- [Derived] Panes J, Louis E, Bossuyt P, Joshi N, Lee WJ, Lacerda AP, Kligys K, Xuan S, Shukla N, Loftus EV Jr. Induction of Endoscopic Response, Remission, and Ulcer-Free Endoscopy With Upadacitinib Is Associated With Improved Clinical Outcomes and Quality of Life in Patients With Crohn's Disease. Inflamm Bowel Dis. 2025 Feb 6;31(2):394-403. doi: 10.1093/ibd/izae200. PMID 39231444
- [Derived] Ghosh S, Feagan BG, Parra RS, Lopes S, Steinlauf A, Kakuta Y, Joshi N, Lee WJ, Lacerda AP, Zhou Q, Xuan S, Kligys K, Shukla N, Louis E. Impact of Upadacitinib Induction and Maintenance Therapy on Health-related Quality of Life, Fatigue, and Work Productivity in Patients with Moderately-to-severely Active Crohn's Disease. J Crohns Colitis. 2024 Nov 4;18(11):1804-1818. doi: 10.1093/ecco-jcc/jjae083. PMID 38835235
- [Derived] Peyrin-Biroulet L, Panaccione R, Louis E, Atreya R, Rubin DT, Lindsay JO, Siffledeen J, Lukin DJ, Wright J, Watanabe K, Ford S, Remple VP, Lacerda AP, Dubcenco E, Garrison A, Zhou Q, Berg S, Anyanwu SI, Schreiber S. Upadacitinib Achieves Clinical and Endoscopic Outcomes in Crohn's Disease Regardless of Prior Biologic Exposure. Clin Gastroenterol Hepatol. 2024 Oct;22(10):2096-2106. doi: 10.1016/j.cgh.2024.02.026. Epub 2024 Mar 15. PMID 38492904
- [Derived] Colombel JF, Hisamatsu T, Atreya R, Bresso F, Thin L, Panaccione R, Parra RS, Ford S, Remple VP, Lacerda AP, Anyanwu SI, Mallick M, Garrison A, Regueiro M. Upadacitinib Reduces Crohn's Disease Symptoms Within the First Week of Induction Therapy. Clin Gastroenterol Hepatol. 2024 Aug;22(8):1668-1677. doi: 10.1016/j.cgh.2024.02.027. Epub 2024 Mar 15. PMID 38492903
- [Derived] Loftus EV Jr, Panes J, Lacerda AP, Peyrin-Biroulet L, D'Haens G, Panaccione R, Reinisch W, Louis E, Chen M, Nakase H, Begun J, Boland BS, Phillips C, Mohamed MF, Liu J, Geng Z, Feng T, Dubcenco E, Colombel JF. Upadacitinib Induction and Maintenance Therapy for Crohn's Disease. N Engl J Med. 2023 May 25;388(21):1966-1980. doi: 10.1056/NEJMoa2212728. PMID 37224198
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants with moderately to severely active Crohn's disease (CD) were randomized at 209 sites in 42 countries. The study consisted of a 12-week double-blind induction treatment period, and a 12-week extended treatment period for participants who did not achieve clinical response at the end of the induction treatment period.
Pre-assignment Details: In Part 1 participants were randomly assigned in a 2:1 ratio to receive upadacitinib 45 mg or placebo, with randomization stratified by Baseline corticosteroid use (yes or no), endoscopic disease severity (Simple Endoscopic Score for Crohn's disease [SES-CD] < 15 and ≥ 15), and the number of previously failed biologic therapies (0, 1, and >1).
Groups:
- Part 1: Placebo: Participants received placebo once daily for 12 weeks in Part 1.
- Part 1: Upadacitinib 45 mg: Participants received 45 mg upadacitinib once daily for 12 weeks in Part 1.
- Part 2: Placebo / Upadacitinib 45 mg: Participants who received placebo during Part 1 and did not achieve clinical response at Week 12 received induction treatment with 45 mg upadacitinib once daily from Week 12 to Week 24.
- Part 2: Upadacitinib 45 mg / Upadacitinib 30 mg: Participants who received upadacitinib during Part 1 and did not achieve clinical response at Week 12 received 30 mg upadacitinib once daily from Week 12 to Week 24.
Period: Part 1: Induction Period (Weeks 1-12)
Arm/Group | Part 1: Placebo | Part 1: Upadacitinib 45 mg | Part 2: Placebo / Upadacitinib 45 mg | Part 2: Upadacitinib 45 mg / Upadacitinib 30 mg
Started | 176 | 350 | 0 | 0
Received Study Drug | 176 | 350 | 0 | 0
Completed | 154 | 330 | 0 | 0
Not Completed | 22 | 20 | 0 | 0
Not completed — Adverse Event | 8 | 12 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 8 | 3 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0
Period: Part 2: Extended Treatment (Weeks 12-24)
Arm/Group | Part 1: Placebo | Part 1: Upadacitinib 45 mg | Part 2: Placebo / Upadacitinib 45 mg | Part 2: Upadacitinib 45 mg / Upadacitinib 30 mg
Started (Participants who were clinical non-responders at the end of the induction period (Week 12) could enter Part 2.) | 0 | 0 | 57 | 59
Completed | 0 | 0 | 49 | 49
Not Completed | 0 | 0 | 8 | 10
Not completed — Adverse Event | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 5
Not completed — Coronavirus Disease-2019 (COVID-19) Infection | 0 | 0 | 0 | 1
Not completed — COVID-19 Logistical Restrictions | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population for the 12-week double-blind induction period includes all randomized participants who received at least one dose of double-blind study drug during Part 1.
Groups:
- Placebo: Participants received placebo once daily for 12 weeks in Part 1.
- Upadacitinib 45 mg: Participants received 45 mg upadacitinib once daily for 12 weeks in Part 1.
- Total: Total of all reporting groups
Arm/Group | Placebo | Upadacitinib 45 mg | Total
Number analyzed (Participants) | 176 | 350 | 526
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (13.63) | 39.7 (13.71) | 39.6 (13.67)
Age, Customized [Count of Participants; unit: Participants]
  18 years - < 40 years | 91 | 193 | 284
  40 years - < 65 years | 80 | 142 | 222
  ≥ 65 years | 5 | 15 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 161 | 243
  Male | 94 | 189 | 283
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 27 | 35
  Not Hispanic or Latino | 168 | 323 | 491
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 36 | 73 | 109
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 17 | 21
  White | 130 | 258 | 388
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Baseline Corticosteroid Use [Count of Participants; unit: Participants]
  Yes | 64 | 126 | 190
  No | 112 | 224 | 336
Number of Previously Failed Biologics [Count of Participants; unit: Participants] — Zero previously failed biologics includes those who never used biologics previously, and/or who have used and stopped due to reasons other than inadequate response and/or intolerance.
  Failed treatment includes an inadequate response or intolerance to treatment.
  Participants
    Zero | 98 | 189 | 287
    One | 28 | 58 | 86
    More than one | 50 | 103 | 153
Endoscopic Disease Severity [Count of Participants; unit: Participants] — Endoscopic disease severity was scored using the Simplified Endoscopic Score for Crohn's Disease (SES-CD). The SES-CD evaluates 4 endoscopic variables (ulcer size, ulcerated surface, affected surface, and narrowing, each on a scale from 0 (none) to 3 (worst) in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, sigmoid and left colon, and rectum). The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores indicate more severe disease.
  Participants
    SES-CD < 15 | 110 | 218 | 328
    SES-CD ≥ 15 | 66 | 132 | 198
Duration of Crohn's Disease [Mean (Standard Deviation); unit: years] | 8.1005 (7.9901) | 9.2993 (9.4684) | 8.8982 (9.0110)
Crohn's Disease Activity Index (CDAI) Score [Mean (Standard Deviation); unit: score on a scale] — The Crohn's Disease Activity Index (CDAI) is a composite instrument that includes participant symptoms evaluated over 7 days (abdominal pain, stool frequency and general well-being), as well as physical and laboratory findings. These items are scored individually, weighted, and do not contribute equally to the overall score. The CDAI is derived from summing up the weighted individual scores of eight items. CDAI approximately ranges from 0 to 600 with higher scores indicating more severe disease. Population: Participants with available data
  score on a scale
    number analyzed (Participants) | 176 | 349 | 525
    (all) | 293.85 (85.378) | 292.42 (81.250) | 292.90 (82.578)
Average Daily Abdominal Pain Score [Mean (Standard Deviation); unit: score on a scale] — Participants were asked to rate their abdominal pain on a daily basis in an electronic diary using the following scale:
  0 = none, 1 = mild, 2 = moderate, 3 = severe.
  The average daily abdominal pain score was calculated using the 4-7 most recent useable days of patient-report outcomes (i.e., excluding days with missing entries or associated with endoscopy procedures) out of the last 14 days prior to the Baseline visit.
  score on a scale | 1.9064 (0.6942) | 1.8917 (0.6795) | 1.8966 (0.6839)
Average Daily Very Soft or Liquid Stool Frequency [Mean (Standard Deviation); unit: stools/day] — Participants were asked to record the number of very soft or liquid stools on a daily basis in an electronic diary.
  The average daily very soft or liquid stool frequency was calculated using the 4-7 most recent useable days of patient-report outcomes (i.e., excluding days with missing entries or associated with endoscopy procedures) out of the last 14 days prior to the Baseline visit.
  stools/day | 5.0857 (2.8366) | 5.1864 (2.6130) | 5.1527 (2.6876)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Remission Per Crohn's Disease Activity Index (CDAI) at Week 12
Description: The co-primary endpoint for United States (US)/Food and Drug Administration (FDA) regulatory purposes was clinical remission based on CDAI at Week 12.
  CDAI is a composite instrument that includes participant symptoms evaluated over 7 days (abdominal pain, stool frequency and general well-being), as well as presence of complications (arthritis/arthralgia, iritis/uveitis, erythema nodosum/pyoderma gangrenosum/aphthous stomatitis, anal fissure/fistula/abscess, other fistula, and fever), the use of antidiarrheal medicines, presence of an abdominal mass, hematocrit, and body weight. These items are scored individually, weighted, and do not contribute equally to the overall score. The CDAI is derived from summing up the weighted individual scores of eight items. CDAI approximately ranges from 0 to 600 with higher scores indicating more severe disease. Clinical remission is defined as a CDAI score less than 150.
Time Frame: Week 12
Population: Randomized participants who received at least one dose of double-blind study drug during Part 1 (intention-to-treat population). Participants with missing data or who withdrew prior to Week 12 were counted as non-responders (non-responder imputation); missing data due to COVID-19 infection or logistical restriction were handled by multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Upadacitinib 45 mg QD: Participants received 45 mg upadacitinib once daily (QD) for 12 weeks in Part 1.
Arm/Group | Placebo | Upadacitinib 45 mg QD
Number analyzed (Participants) | 176 | 350
percentage of participants | 29.1 [22.4 to 35.8] | 49.5 [44.2 to 54.8]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 45 mg QD; Comparison of the upadacitinib group and placebo group was performed using the Cochran Mantel-Haenszel (CMH) test adjusting for stratification factors (baseline steroid use [Yes, No], endoscopic disease severity [SES-CD < 15, ≥ 15] and number of prior biologics with prior inadequate response or intolerance [0, 1, > 1]); Test type: Superiority — The overall type I error rate of the co-primary and ranked secondary endpoints were strongly controlled using a fixed sequence multiple-testing procedure as well as a Holm procedure. The testing utilized the sequence of hypothesis testing for the co-primary endpoints using two-sided α of 0.05 followed by a set of ranked key secondary endpoints, defined separately for US/FDA and European Union/European Medicines Agency regulatory purposes; p < 0.0001, Cochran-Mantel-Haenszel; Cochran Mantel-Haenszel test adjusted for stratification factors; Adjusted Response Rate Difference = 20.8, 95% CI 2-sided [12.7 to 28.8] — Adjusted response rate difference (Upadacitinib - Placebo) calculated based on CMH test adjusted for stratification factors

2. Primary Outcome: Percentage of Participants With Clinical Remission Per Patient-Reported Outcomes (PROs) at Week 12
Description: The co-primary endpoint for European Union (EU)/European Medicines Agency (EMA) regulatory purposes was clinical remission defined based on two patient reported outcomes, average daily stool frequency (SF) and average daily abdominal pain score (APS). Clinical remission per PROs was defined as average daily very soft or liquid SF ≤ 2.8 and average daily APS ≤ 1.0 and neither worse than Baseline.
  Participants recorded APS and the number of very soft or liquid SF daily in an electronic diary. Abdominal pain was rated on a scale from 0 (none) to 3 (severe).
  The average daily very soft or liquid SF and APS were calculated using the 4-7 most recent useable days of patient-report outcomes (i.e., excluding days with missing entries or associated with endoscopy procedures) out of the last 14 days prior to the Week 12 visit.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 45 mg QD
Number analyzed (Participants) | 176 | 350
percentage of participants | 22.2 [16.0 to 28.3] | 50.7 [45.5 to 56.0]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 45 mg QD; Test type: Superiority — The overall type I error rate of the co-primary and ranked secondary endpoints were strongly controlled using a fixed sequence multiple-testing procedure as well as a Holm procedure. The testing utilized the sequence of hypothesis testing for the co-primary endpoints using two-sided α of 0.05 followed by a set of ranked key secondary endpoints, defined separately for US/FDA and EU/EMA regulatory purposes; p < 0.0001, Cochran-Mantel-Haenszel; Cochran Mantel-Haenszel test adjusted for stratification factors; Adjusted Response Rate Difference = 28.7, 95% CI 2-sided [20.9 to 36.4] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Percentage of Participants With Endoscopic Response at Week 12
Description: Endoscopic response at Week 12 was a co-primary endpoint for both the US/FDA and EU/EMA regulatory purposes. Endoscopic response was defined as greater than 50% decrease in Simple Endoscopic Score for Crohn's Disease (SES-CD) from Baseline of the induction study (or for participants with an SES-CD of 4 at Baseline, at least a 2-point reduction from Baseline), as scored by independent external and blinded central readers.
  The SES-CD evaluates 4 endoscopic variables (ulcer size, ulcerated surface, affected surface, and narrowing, each on a scale from 0 (none) to 3 in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, sigmoid and left colon, and rectum). The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores indicate more severe disease.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 45 mg QD
Number analyzed (Participants) | 176 | 350
percentage of participants | 13.1 [8.1 to 18.0] | 45.5 [40.3 to 50.8]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 45 mg QD; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran Mantel-Haenszel test adjusted for stratification factors; Adjusted Response Rate Difference = 33.0, 95% CI 2-sided [26.2 to 39.9] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants With Endoscopic Remission at Week 12
Description: Endoscopic remission is defined as an SES-CD ≤ 4 and at least 2 point reduction from Baseline and no subscore > 1 in any individual variable,as scored by independent external and blinded central readers.
  The SES-CD evaluates 4 endoscopic variables (ulcer size, ulcerated surface, affected surface, and narrowing, each on a scale from 0 (none) to 3 in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, sigmoid and left colon, and rectum). The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores indicate more severe disease.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 45 mg QD
Number analyzed (Participants) | 176 | 350
percentage of participants | 7.4 [3.5 to 11.3] | 28.9 [24.2 to 33.7]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 45 mg QD; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran Mantel-Haenszel test adjusted for stratification factors; Adjusted Response Rate Difference = 21.8, 95% CI 2-sided [15.8 to 27.8] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants Who Discontinued Corticosteroid Use for Crohn's Disease and Achieved Clinical Remission Per CDAI at Week 12
Description: Corticosteroid-free clinical remission is defined as participants who discontinued corticosteroid use for CD and achieved clinical remission per CDAI at Week 12, assessed for participants taking corticosteroids for CD at Baseline.
  CDAI is a composite instrument that includes participant symptoms evaluated over 7 days (abdominal pain, stool frequency and general well-being), as well as presence of complications (arthritis/arthralgia, iritis/uveitis, erythema nodosum/pyoderma gangrenosum/aphthous stomatitis, anal fissure/fistula/abscess, other fistula, and fever), the use of antidiarrheal medicines, presence of an abdominal mass, hematocrit, and body weight. These items are scored individually, weighted, and do not contribute equally to the overall score. The CDAI is derived from summing up the weighted individual scores of eight items. CDAI approximately ranges from 0 to 600 with higher scores indicating more severe disease. Clinical remission is defined as CDAI score less than 150.
Time Frame: Week 12
Population: Randomized participants who received at least one dose of double-blind study drug during Part 1 (intention-to-treat population) who were taking corticosteroids for Crohn's disease at Baseline.
  Participants with missing data or who withdrew prior to Week 12 were counted as non-responders (non-responder imputation); missing data due to COVID-19 infection or logistical restriction were handled by multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 45 mg QD
Number analyzed (Participants) | 64 | 126
percentage of participants | 15.7 [6.8 to 24.7] | 42.9 [34.2 to 51.5]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 45 mg QD; Test type: Superiority — The overall type I error rate of the co-primary and ranked secondary endpoints were strongly controlled using a fixed sequence multiple-testing procedure as well as a Holm procedure. The testing utilized the sequence of hypothesis testing for the co-primary endpoints using two-sided α of 0.05 followed by a set of ranked key secondary endpoints. This endpoint was a ranked key secondary endpoint for US/FDA regulatory purposes; p < 0.0001, Cochran-Mantel-Haenszel; Cochran Mantel-Haenszel test adjusted for stratification factors endoscopic disease severity and number of prior failed biologic therapies; Adjusted Response Rate Difference = 27.7, 95% CI 2-sided [15.7 to 39.8] — Adjusted response rate difference (Upadacitinib - Placebo) calculated based on CMH test adjusted for stratification factors endoscopic disease severity and number of prior biologic failed

6. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) at Week 12
Description: The FACIT-Fatigue questionnaire is a self-administered patient questionnaire that consists of 13 questions designed to measure the degree of fatigue experienced by participants in the previous 7 days, including physical fatigue (e.g., I feel tired), functional fatigue (e.g., trouble finishing things), emotional fatigue (e.g., frustration), and social consequences of fatigue (e.g., limits social activity). Participants respond to the questions on a scale from 0 (not at all) to 4 (very much). The FACIT-Fatigue score is computed by summing the item scores, after reversing those items that are worded in the negative direction. The FACIT-Fatigue score ranges from 0 to 52, where higher scores represent less fatigue. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: Randomized participants who received at least one dose of double-blind study drug during Part 1 (intention-to-treat population); missing data were handled using a mixed-effect model with repeated measurements (MMRM). The Overall Number of Participants Analyzed presented below is based on the number of participants with non-missing Baseline and Week 12 values.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 45 mg QD
Number analyzed (Participants) | 133 | 304
score on a scale | 5.0 [3.2 to 6.8] | 11.3 [10.0 to 12.5]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 45 mg QD; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Mixed-effect Model Repeated Measurement; MMRM model with fixed effects of treatment, visit, and treatment-by-visit interaction, stratification factors, and Baseline value as covariate; Least Squares (LS) Mean Difference = 6.3, 95% CI 2-sided [4.2 to 8.3], Standard Error of Mean 1.05

7. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Week 12
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) is used to assess health-related quality of life (HRQoL) in patients with inflammatory bowel disease. It consists of 32 questions evaluating bowel and systemic symptoms, as well as emotional and social functions. Each question is answered on a scale from 1 (worst) to 7 (best). The total score ranges from 32 to 224 with higher scores indicating better health-related quality of life. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Upadacitinib 45 mg QD
Number analyzed (Participants) | 134 | 304
score on a scale | 24.423 [19.007 to 29.840] | 46.265 [42.495 to 50.035]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 45 mg QD; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Mixed-effect Model Repeated Measurement; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = 21.842, 95% CI 2-sided [15.566 to 28.118], Standard Error of Mean 3.1933

8. Secondary Outcome: Percentage of Participants Achieving Clinical Response 100 (CR-100) at Week 2
Description: Clinical response 100 (CR-100) is defined as a decrease of at least 100 points in CDAI from Baseline.
  CDAI is a composite instrument that includes participant symptoms evaluated over 7 days (abdominal pain, stool frequency and general well-being), as well as presence of complications (arthritis/arthralgia, iritis/uveitis, erythema nodosum/pyoderma gangrenosum/aphthous stomatitis, anal fissure/fistula/abscess, other fistula, and fever), the use of antidiarrheal medicines, presence of an abdominal mass, hematocrit, and body weight. These items are scored individually, weighted, and do not contribute equally to the overall score. The CDAI is derived from summing up the weighted individual scores of eight items. CDAI approximately ranges from 0 to 600 with higher scores indicating more severe disease.
Time Frame: Baseline and Week 2
Population: Randomized participants who received at least one dose of double-blind study drug during Part 1 (intention-to-treat population). Participants with missing data or who withdrew prior to Week 2 were counted as non-responders (non-responder imputation); missing data due to COVID-19 infection or logistical restriction were handled by multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 45 mg QD
Number analyzed (Participants) | 176 | 350
percentage of participants | 20.4 [14.4 to 26.5] | 32.2 [27.3 to 37.1]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 45 mg QD; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0022, Cochran-Mantel-Haenszel; Cochran Mantel-Haenszel test adjusted for stratification factors; Adjusted Response Rate Difference = 11.7, 95% CI 2-sided [4.2 to 19.2] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Percentage of Participants Achieving Clinical Response 100 (CR-100) at Week 12
Description: as for outcome 8
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 45 mg QD
Number analyzed (Participants) | 176 | 350
percentage of participants | 37.3 [30.1 to 44.5] | 56.6 [51.4 to 61.8]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 45 mg QD; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran Mantel-Haenszel test adjusted for stratification factors; Adjusted Response Rate Difference = 19.8, 95% CI 2-sided [11.3 to 28.4] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Percentage of Participants With Clinical Remission Per CDAI at Week 4
Description: CDAI is a composite instrument that includes participant symptoms evaluated over 7 days (abdominal pain, stool frequency and general well-being), as well as presence of complications (arthritis/arthralgia, iritis/uveitis, erythema nodosum/pyoderma gangrenosum/aphthous stomatitis, anal fissure/fistula/abscess, other fistula, and fever), the use of antidiarrheal medicines, presence of an abdominal mass, hematocrit, and body weight. These items are scored individually, weighted, and do not contribute equally to the overall score. The CDAI is derived from summing up the weighted individual scores of eight items. CDAI approximately ranges from 0 to 600 with higher scores indicating more severe disease. Clinical remission is defined as CDAI score less than 150.
Time Frame: Week 4
Population: Randomized participants who received at least one dose of double-blind study drug during Part 1 (intention-to-treat population). Participants with missing data or who withdrew prior to Week 4 were counted as non-responders (non-responder imputation); missing data due to COVID-19 infection or logistical restriction were handled by multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 45 mg QD
Number analyzed (Participants) | 176 | 350
percentage of participants | 26.7 [20.2 to 33.3] | 37.1 [32.1 to 42.2]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 45 mg QD; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0071, Cochran-Mantel-Haenszel; Cochran Mantel-Haenszel test adjusted for stratification factors; Adjusted Response Rate Difference = 10.8, 95% CI 2-sided [2.9 to 18.6] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Percentage of Participants With Hospitalizations Due to Crohn's Disease (CD) During the 12-Week Induction Period
Description: This was assessed by reviewing participant's hospitalization data.
Time Frame: 12 weeks
Population: Randomized participants who received at least one dose of double-blind study drug during Part 1 (intention-to-treat population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 45 mg QD
Number analyzed (Participants) | 176 | 350
percentage of participants | 5.1 [1.9 to 8.4] | 3.7 [1.7 to 5.7]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 45 mg QD; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.4494, Chi-squared; Response Rate Difference = -1.4, 95% CI 2-sided [-5.2 to 2.4] — Response rate difference = Upadacitinib - Placebo

12. Secondary Outcome: Percentage of Participants With Resolution of Extra-Intestinal Manifestation (EIMs) at Week 12
Description: EIMs are defined as manifestations of Crohn's disease in areas of the body other than the digestive tract, including eyes, skin, joints, mouth, and liver.
  Only participants with any EIM present at Baseline were included in the analysis of resolution of EIMs. Resolution of EIMs was defined as absence of all EIMs at the Week 12 visit.
Time Frame: Week 12
Population: Randomized participants who received at least one dose of double-blind study drug during Part 1 (intention-to-treat population) with any EIM at Baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 45 mg QD
Number analyzed (Participants) | 78 | 151
percentage of participants | 20.9 [11.8 to 30.1] | 28.5 [21.3 to 35.7]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 45 mg QD; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.1044, Cochran-Mantel-Haenszel; Cochran Mantel-Haenszel test adjusted for stratification factors; Adjusted Response Rate Difference = 9.0, 95% CI 2-sided [-1.9 to 19.9] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Percentage of Participants With Clinical Remission Per PROs at Week 4
Description: Clinical remission per PROs was defined as average daily very soft or liquid SF ≤ 2.8 and average daily APS ≤ 1.0 and neither worse than Baseline.
  Participants recorded APS and the number of liquid or very soft SF daily in an electronic diary. Abdominal pain was rated on a scale from 0 (none) to 3 (severe).
  The average daily very soft or liquid SF and APS were calculated using the 4-7 most recent useable days of patient-reported outcomes (i.e., excluding days with missing entries or associated with endoscopy procedures) out of the last 14 days prior to the Week 4 visit.
Time Frame: Week 4
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 45 mg QD
Number analyzed (Participants) | 176 | 350
percentage of participants | 14.8 [9.5 to 20.0] | 35.7 [30.7 to 40.7]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 45 mg QD; Test type: Superiority — The overall type I error rate of the co-primary and ranked secondary endpoints were strongly controlled using a fixed sequence multiple-testing procedure as well as a Holm procedure. The testing utilized the sequence of hypothesis testing for the co-primary endpoints using two-sided α of 0.05 followed by a set of ranked key secondary endpoints. This endpoint was a ranked key secondary endpoint for EU/EMA regulatory purposes; p < 0.0001, Cochran-Mantel-Haenszel; Cochran Mantel-Haenszel test adjusted for stratification factors; Adjusted Response Rate Difference = 21.2, 95% CI 2-sided [14.3 to 28.2] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Percentage of Participants Who Discontinued Corticosteroid Use for Crohn's Disease and Achieved Clinical Remission Per PROs at Week 12
Description: Corticosteroid-free clinical remission is defined as participants who discontinued corticosteroid use for CD and achieved clinical remission per PROs at Week 12, assessed for participants taking corticosteroids for CD at Baseline.
  Clinical remission per PROs was defined as average daily very soft or liquid stool frequency (SF) ≤ 2.8 and average daily APS ≤ 1.0 and neither worse than Baseline.
  Participants recorded APS and the number of liquid or very soft SF daily in an electronic diary. Abdominal pain was rated on a scale from 0 (none) to 3 (severe).
  The average daily liquid or very soft SF and APS were calculated using the 4-7 most recent useable days of patient-reported outcomes (i.e., excluding days with missing entries or associated with endoscopy procedures) out of the last 14 days prior to the Week 12 visit.
Time Frame: Week 12
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 45 mg QD
Number analyzed (Participants) | 64 | 126
percentage of participants | 12.5 [4.4 to 20.6] | 44.4 [35.8 to 53.1]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 45 mg QD; Test type: Superiority — [test comment as in outcome 13, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran Mantel-Haenszel test adjusted for stratification factors; Adjusted Response Rate Difference = 32.6, 95% CI 2-sided [21.5 to 43.7] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Part 1: 12 weeks Part 2: 12 weeks
Arm/Group | Part 1: Placebo | Part 1: Upadacitinib 45 mg | Part 2: Placebo / Upadacitinib 45 mg | Part 2: Upadacitinib 45 mg / Upadacitinib 30 mg
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/350 | 0/57 | 1/59
Serious Adverse Events (participants affected / at risk) | 12/176 | 24/350 | 4/57 | 6/59
Other Adverse Events (participants affected / at risk) | 37/176 | 92/350 | 14/57 | 13/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (N=176) | Part 1: Upadacitinib 45 mg (N=350) | Part 2: Placebo / Upadacitinib 45 mg (N=57) | Part 2: Upadacitinib 45 mg / Upadacitinib 30 mg (N=59)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 5 (5) | 7 (8) | 1 (1) | 2 (2)
ENTERITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ILEAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS ROTAVIRUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RECTAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
METASTATIC CUTANEOUS CROHN'S DISEASE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (N=176) | Part 1: Upadacitinib 45 mg (N=350) | Part 2: Placebo / Upadacitinib 45 mg (N=57) | Part 2: Upadacitinib 45 mg / Upadacitinib 30 mg (N=59)
ANAEMIA (Blood and lymphatic system disorders) | 8 (8) | 21 (23) | 3 (3) | 2 (2)
CROHN'S DISEASE (Gastrointestinal disorders) | 13 (13) | 5 (5) | 1 (1) | 3 (3)
PYREXIA (General disorders) | 2 (2) | 14 (15) | 1 (1) | 3 (3)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 6 (6) | 16 (16) | 2 (2) | 4 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 (9) | 9 (10) | 3 (3) | 1 (1)
ACNE (Skin and subcutaneous tissue disorders) | 1 (1) | 24 (24) | 3 (3) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 4 (4) | 13 (14) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT03345849/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT03345849/SAP_002.pdf